CLINICAL TRIAL: NCT01266330
Title: Dairy Attenuation of Oxidative and Inflammatory Stress in Metabolic Syndrome
Brief Title: Dairy Attenuation of Metabolic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Michael B. Zemel, The University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R011770040
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Oxidative Stress; Inflammation
Keywords: dairy; inflammation; reactive oxygen species; oxidative stress; body composition
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dairy (Active Comparator): <0.5 standard dairy servings/day
  Interventions: Dietary Supplement: Low Dairy
- Adequate dairy (Experimental): 3.5 standard dairy servings per day
  Interventions: Dietary Supplement: Adequate Dairy

INTERVENTIONS:
Dietary Supplement: Low Dairy — Less than 0.5 standard servings of dairy products per day
  Arms: Low Dairy
Dietary Supplement: Adequate Dairy — 3.5 standard servings of dairy foods per day
  Arms: Adequate dairy

SUMMARY:
Forty overweight and obese subjects (BMI 25-39.9) with metabolic syndrome will be randomized to inadequate dairy (<0.5 serving/day) and adequate dairy (3.5 servings/day) weight maintenance (eucaloric) diets for 12 weeks. Body weight will be measured weekly and body composition (via dual X-ray absorptiometry), insulin sensitivity index, plasma lipids and calcitrophic hormones will be measured at weeks 0, 4 and 12 of the dietary intervention. Oxidative burden will be assessed by measurement of plasma malonaldehyde, 8-isoprostane F2α and oxidized LDL and inflammatory stress will be assessed by measurement of IL-6, IL-15, MCP, C-reactive protein, adiponectin and TNF-α levels in plasma at 0, 1, 4 and 12 weeks). An additional global evaluation of diet-induced changes in cytokines will be conducted using cytokine protein arrays to profile relative changes in 36 additional potentially relevant cytokines. All data will be analyzed via two-factor (diet X obesity status) multivariate analysis of variance (MANOVA)

DETAILED DESCRIPTION:
This study is designed to determine the effects of a dairy-rich diet on oxidative and inflammatory stress in metabolic syndrome patients in the presence and absence of obesity. Forty overweight and obese subjects (BMI 25-39.9) with metabolic syndrome as defined by NCEP ATP III criteria will be randomized to inadequate (0-0.5 daily serving) or adequate (3.5 servings) dairy diets in the presence of a eucaloric weight maintenance diet for 12 weeks. All subjects will undergo a 14-day lead-in period to establish a stable baseline of dietary and physiological measures (described below), followed by the 12-week intervention period. Baseline dietary assessments will be conducted by the project dietitian during the two-week lead-in period which will be used to provide an initial estimate of a maintenance level of caloric intake. This will be refined by calculating energy needs using DRI equations for calculation of age- and physical activity (PA) adjusted total energy expenditure (TEE) for men and women. Energy requirements will be confirmed via measurement of resting metabolic rate via indirect calorimetry.

Subjects will be given diets isocaloric to those consumed during the lead-in period, with macronutrient and fiber levels maintained equivalent at levels approximating the estimated U.S. average (described in Diets section). Subjects on the inadequate dairy diets will be assigned diets containing < 600 mg Ca/day and <0.5 daily serving of dairy foods, and subjects on the adequate dairy diets will be assigned diets containing 1200 - 1400 mg Ca/day and 3.5 daily servings of dairy (milk, yogurt, hard cheese). Two of the three dairy servings consumed daily by those on the high dairy diet will be milk and/or yogurt to ensure sufficient consumption of whey proteins. All subjects will be provided individual instruction, counseling and assessment from the study dietitian regarding dietary adherence and the development and reinforcement of strategies for continued success, and diets will be monitored weekly. Physical activity will be assessed using pedometer counts and maintained at approximately pre-study levels throughout the study. Pedometer counts will be recorded daily for the 14-day lead-in period and the value averaged to provide a pre-study baseline. Subjects will be asked to maintain the same level of activity (plus or minus 500 steps/day) and will use pedometers for self-assessment. Pedometer counts will be recorded and provided to the study staff on a weekly basis, along with the diet records.

Body weight, waist circumference, and blood pressure will be measured weekly and body composition (via dual X-ray absorptiometry) will be measured at weeks 0, 4 and 12 of the dietary intervention. Resting metabolic rate and respiratory quotient will be assessed at weeks 0 and 12. Oxidative burden will be assessed by measurement of plasma malonaldehyde, 8-isoprostane F2α and oxidized LDL at weeks 0, 1, 4 and 12, and inflammatory stress will be assessed by measurement of IL-6, IL-15, MCP, C-reactive protein, adiponectin and TNF-α levels in plasma at the same time intervals. Glucose tolerance, HOMAIR, fasting plasma lipids, PTH and 1,25-(OH)2-D levels will be determined at the same time intervals (0, 4, and 12 weeks). All data will be analyzed via two-factor multivariate analysis of variance (MANOVA).

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of metabolic syndrome as defined by NCEP ATP III criteria: Presence of three or more of the following risk determinants:

  * Abdominal obesity (This criterion must be met by all obese subjects entered into the study)

    * Waist circumference >102 cm for males
    * Waist circumference >88 cm for females
  * Triglycerides >150 mg/dL
  * HDL cholesterol <40 mg/dL (men); < 50 mg/dL (women)
  * Blood pressure >130/>85 mm Hg (This criterion must be met by all subjects [overweight and obese] entered into the study).
  * Fasting glucose >100 mg/dL

    * Body mass index (BMI) 25-39.9
    * Age 18-50 years
    * Weight stable: no more than 1 kg weight gain or loss during past four weeks

Exclusion Criteria:

* • BMI < 25 or >40

  * Type II diabetes requiring the use of any oral antidiabetic agent and/or insulin (because of confounding effects on ROS)
  * Adverse response to study foods (lactose intolerance, dairy intolerance, dairy allergy); this will be determined by self-report.
  * history or presence of significant metabolic disease which could impact on the results of the study (i.e. endocrine, hepatic, renal disease)
  * history of eating disorder
  * presence of active gastrointestinal disorders such as malabsorption syndromes
  * pregnancy or lactation
  * use of obesity pharmacotherapeutic agents within the last 6 months
  * use of over-the-counter anti-obesity agents (e.g. those containing phenylpropanalamine, ephedrine and/or caffeine) within the last 3 months
  * Chronic use of anti-inflammatory agents within the last four weeks
  * Use of antioxidant supplements within the last four weeks
  * Recent (current or past 12 weeks) use of any psychotropic medication
  * Recent (past four weeks) initiation of an exercise program
  * Recent (past twelve weeks) initiation of hormone replacement therapy or change in HRT regimen
  * Recent (past twelve weeks) initiation of hormonal birth control or change in hormonal birth control regimen
  * Recent (past 12-weeks) history of tobacco use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
Body composition | 12 weeks
  DEXA assessment
Oxidative Stress | 12 weeks
  plasma malonaldehyde, 8-isoprostane F2α and oxidized LDL
Inflammatory stress | 12 weeks
  Plasma L-6, IL-15, MCP, C-reactive protein, adiponectin and TNF-α

SECONDARY OUTCOMES:
Insulin sensitivituy | 12 weeks
  Glucose, insulin and HOMA
Blood pressure | 12 weeks
Lipids | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Zemel, Ph.D., Principal Investigator — The University of Tennessee
Locations (1):
- The University of Tennessee Nutrition and Metabolic Research Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Stancliffe RA, Thorpe T, Zemel MB. Dairy attentuates oxidative and inflammatory stress in metabolic syndrome. Am J Clin Nutr. 2011 Aug;94(2):422-30. doi: 10.3945/ajcn.111.013342. Epub 2011 Jun 29. PMID 21715516